CLINICAL TRIAL: NCT06772597
Title: A Phase 2 Open-label Study of Setmelanotide in Patients With Prader-Willi Syndrome
Brief Title: A Study of Setmelanotide in Patients With Prader-Willi Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-043
Record Dates: First submitted 2025-01-10; First posted 2025-01-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prader-Willi Syndrome; Obesity; Hyperphagia
Keywords: melanocortin 4 receptor (MC4R), MC4R agonist
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity; Hyperphagia | interventions — setmelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setmelanotide (Open-label) (Experimental)
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — Setmelanotide (daily subcutaneous injection)
  Other Names: Imcivree

SUMMARY:
This is a Phase 2, open-label study designed to assess the safety and efficacy of setmelanotide in patients with obesity due to Prader-Willi Syndrome (PWS) who are 6 to 65 years of age. Up to 20 patients are planned to be enrolled. Patients will take a daily subcutaneous dose of open-label setmelanotide for up to 52 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of Prader-Willi Syndrome (PWS)
* Age 6 to 65
* BMI ≥30 kg/m2 for patients ≥18 years of age or BMI ≥95th Percentile for age and sex
* Agree to use a highly effective form of contraception and follow the study contraception requirements throughout study duration and for 90 days after.
* Patient and/or guardian is able to communicate well with the Investigator, understand and comply with the requirements of the study, and understand English and sign the written informed consent.

Exclusion Criteria:

* Use of weight modulating medications
* Abnormal eGFR, ALT, AST, and bilirubin values
* Current, clinically significant pulmonary, cardiac, metabolic, or oncologic disease considered severe enough to interfere with the trial and/or confound the results.
* Participation in any clinical trial with an investigational drug/device within 3 months or 5 half-lives, whichever is longer, prior to the first trial dose
* Hypersensitivity to setmelanotide
* Diagnosis of severe psychiatric disorders
* Pregnant and/or breastfeeding

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) | Baseline to Week 52

SECONDARY OUTCOMES:
Proportion of patients who achieve 5% reduction in BMI | Baseline to Week 52
Mean percent change in BMI | Baseline to Week 52
Mean percent change in BMI and weight in patients ≥18 years of age | Baseline to Week 52
Mean change in BMI Z-Score and BMI % of 95th percentile | Baseline to Week 52
Proportion of patients who achieved 5% reduction in weight from Baseline in patients ≥18 years of age and who achieved ≥0.2 reduction in BMI Z-score in patients <18 years of age | Baseline to Week 52
Mean change in the weekly average of the Prader-Willi Syndrome Food Problem Diary (PWS-FPD) total score | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (1):
- University of Florida, Gainesville, Florida, United States